CLINICAL TRIAL: NCT03392610
Title: Reusable Flexible Bronchoscopes Versus Single Use Bronchoscopes : a Satisfaction Survey
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: I17023
Record Dates: First submitted 2017-12-06; First posted 2018-01-08 (Actual); Last update posted 2018-07-09 (Actual); Status verified 2017-10

CONDITIONS: Bronchoscope Users
Keywords: Intratracheal intubation, bronchoscopy, bronchoalveolar lavage, endoscopy, pulmonary medicine, critical care, anesthesia department, disinfection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Bronchial endoscopy: Compare quality procedures performed with reusable versus disposable bronchoscopes in respiratory endoscopy unit
- Critical care unit: Compare quality procedures performed with reusable versus disposable bronchoscopes in critical care unit
- Anesthesia department: Compare quality procedures performed with reusable versus disposable bronchoscopes in anesthesia department

SUMMARY:
Reusable (RU) flexible bronchoscopes (FB) require intermediate level disinfection operations to prevent transmission of infectious agents from patient to patient. These operations have a significant material and human cost and impact their availability in case of emergency. One alternative is the use of disposable FB.

The aim of the study is to evaluate the quality of FB during procedures carried out with each of the two solutions in intensive care unit (ICU), respiratory endoscopy (RE) and anesthesia (A) department.

A prospective non-interventional and non-randomized monocentric study compare the operator satisfaction of therapeutic procedures performed with RU FB (EB FujifilmTM range, FB/FI PentaxMedicalTM range, StorzTM intubation FB) versus disposable FB (aScope 3® and aScope 4® (AmbuTM), Broncoflex® (AxessvisionTM). An evaluation form is completed by the operator at the end of procedure. Judging criteria, rated from 0 to 10, concern handling, ergonomics, image and suction quality.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent a therapeutic bronchoscopy (Bronchoalveolar lavage, protected bronchial brushing, suction, difficult intubation)
* Patient followed or treated at the Limoges University Hospital

Exclusion Criteria:

* Patient < 18 years
* Diagnostic bronchoscopy
* Interventional bronchoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent therapeutic bronchoscopy in anesthesia department, respiratory endoscopy unit, and critical care unit
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-12-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Bronchoscopes overall reliability: comparison of physician satisfaction scores (rated on a scale from 0 to 10) between RU FB and disposable FB | Time required to carry out the bronchoscopy (between 5 and 15 minutes)
  A score is given per bronchoscopy (RU FB or disposable FB) All scores are aggregated as an average for FB RU and as an average for disposable FBs The 2 averages obtained are compared by a Student T- test after verification of the application conditions by a Fisher F-test (alpha = 5% threshold)
  Additional information about the measurement:
  2/10: poor 4/10: mediocre 6/10: sufficient 8/10: suitable 10/10: excellent

SECONDARY OUTCOMES:
Passage of the endoscope through the probe (intubated patient): comparison of physician satisfaction scores (rated on a scale from 0 to 10) between RU FB and disposable FB | time required to carry out the bronchoscopy (between 5 and 15 minutes)
  A score is given per bronchoscopy (RU FB or disposable FB) All scores are aggregated as an average for FB RU and as an average for disposable FBs The 2 averages obtained are compared by a Student T- test after verification of the application conditions by a Fisher F-test (alpha = 5% threshold)
  Additional information about the measurement:
  2/10: very difficult 4/10: difficult 6/10: relatively easy 8/10: easy 10/10: very easy
Bronchoscope access to trachea (non-intubated patient): comparison of physician satisfaction scores (rated on a scale from 0 to 10) between RU FB and disposable FB | time required to carry out the bronchoscopy (between 5 and 15 minutes)
  A score is given per bronchoscopy (RU FB or disposable FB) All scores are aggregated as an average for FB RU and as an average for disposable FBs The 2 averages obtained are compared by a Student T- test after verification of the application conditions by a Fisher F-test (alpha = 5% threshold)
  Additional information about the measurement:
  2/10: very difficult 4/10: difficult 6/10: relatively easy 8/10: easy 10/10: very easy
Bronchial catheterization: comparison of physician satisfaction scores (rated on a scale from 0 to 10) between RU FB and disposable | time required to carry out the bronchoscopy (between 5 and 15 minutes)
  A score is given per bronchoscopy (RU FB or disposable FB) All scores are aggregated as an average for FB RU and as an average for disposable FBs The 2 averages obtained are compared by a Student T- test after verification of the application conditions by a Fisher F-test (alpha = 5% threshold)
  Additional information about the measurement:
  2/10: very difficult 4/10: difficult 6/10: relatively easy 8/10: easy 10/10: very easy
Left/right rotation of the insertion tube: comparison of physician satisfaction scores (rated on a scale from 0 to 10) between RU FB and disposable FB | time required to carry out the bronchoscopy (between 5 and 15 minutes)
  A score is given per bronchoscopy (RU FB or disposable FB) All scores are aggregated as an average for FB RU and as an average for disposable FBs The 2 averages obtained are compared by a Student T- test after verification of the application conditions by a Fisher F-test (alpha = 5% threshold)
  Additional information about the measurement:
  2/10: poor 4/10: mediocre 6/10: sufficient 8/10: suitable 10/10: excellent
Crutch handling: comparison of physician satisfaction scores (rated on a scale from 0 to 10) between RU FB and disposable FB | time required to carry out the bronchoscopy (between 5 and 15 minutes)
  A score is given per bronchoscopy (RU FB or disposable FB) All scores are aggregated as an average for FB RU and as an average for disposable FBs The 2 averages obtained are compared by a Student T- test after verification of the application conditions by a Fisher F-test (alpha = 5% threshold)
  Additional information about the measurement:
  2/10: poor 4/10: mediocre 6/10: sufficient 8/10: suitable 10/10: excellent
Close brightness: comparison of physician satisfaction scores (rated on a scale from 0 to 10) between RU FB and disposable FB | time required to carry out the bronchoscopy (between 5 and 15 minutes)
  A score is given per bronchoscopy (RU FB or disposable FB) All scores are aggregated as an average for FB RU and as an average for disposable FBs The 2 averages obtained are compared by a Student T- test after verification of the application conditions by a Fisher F-test (alpha = 5% threshold)
  Additional information about the measurement:
  2/10: poor 4/10: mediocre 6/10: sufficient 8/10: suitable 10/10: excellent
Outer brightness: comparison of physician satisfaction scores (rated on a scale from 0 to 10) between RU FB and disposable FB | time required to carry out the bronchoscopy (between 5 and 15 minutes)
  A score is given per bronchoscopy (RU FB or disposable FB) All scores are aggregated as an average for FB RU and as an average for disposable FBs The 2 averages obtained are compared by a Student T- test after verification of the application conditions by a Fisher F-test (alpha = 5% threshold)
  Additional information about the measurement:
  2/10: poor 4/10: mediocre 6/10: sufficient 8/10: suitable 10/10: excellent
Close focus: comparison of physician satisfaction scores (rated on a scale from 0 to 10) between RU FB and disposable FB | time required to carry out the bronchoscopy (between 5 and 15 minutes)
  A score is given per bronchoscopy (RU FB or disposable FB) All scores are aggregated as an average for FB RU and as an average for disposable FBs The 2 averages obtained are compared by a Student T- test after verification of the application conditions by a Fisher F-test (alpha = 5% threshold)
  Additional information about the measurement:
  2/10: poor 4/10: mediocre 6/10: sufficient 8/10: suitable 10/10: excellent
Close sharpness: comparison of physician satisfaction scores (rated on a scale from 0 to 10) between RU FB and disposable | time required to carry out the bronchoscopy (between 5 and 15 minutes)
  A score is given per bronchoscopy (RU FB or disposable FB) All scores are aggregated as an average for FB RU and as an average for disposable FBs The 2 averages obtained are compared by a Student T- test after verification of the application conditions by a Fisher F-test (alpha = 5% threshold)
  Additional information about the measurement:
  2/10: poor 4/10: mediocre 6/10: sufficient 8/10: suitable 10/10: excellent
Outer sharpness: comparison of physician satisfaction scores (rated on a scale from 0 to 10) between RU FB and disposable FB | time required to carry out the bronchoscopy (between 5 and 15 minutes)
  A score is given per bronchoscopy (RU FB or disposable FB) All scores are aggregated as an average for FB RU and as an average for disposable FBs The 2 averages obtained are compared by a Student T- test after verification of the application conditions by a Fisher F-test (alpha = 5% threshold)
  Additional information about the measurement:
  2/10: poor 4/10: mediocre 6/10: sufficient 8/10: suitable 10/10: excellent
Color reproduction: comparison of physician satisfaction scores (rated on a scale from 0 to 10) between RU FB and disposable FB | time required to carry out the bronchoscopy (between 5 and 15 minutes)
  A score is given per bronchoscopy (RU FB or disposable FB) All scores are aggregated as an average for FB RU and as an average for disposable FBs The 2 averages obtained are compared by a Student T- test after verification of the application conditions by a Fisher F-test (alpha = 5% threshold)
  Additional information about the measurement:
  2/10: poor 4/10: mediocre 6/10: sufficient 8/10: suitable 10/10: excellent
Image contrast: comparison of physician satisfaction scores (rated on a scale from 0 to 10) between RU FB and disposable FB | time required to carry out the bronchoscopy (between 5 and 15 minutes)
  A score is given per bronchoscopy (RU FB or disposable FB) All scores are aggregated as an average for FB RU and as an average for disposable FBs The 2 averages obtained are compared by a Student T- test after verification of the application conditions by a Fisher F-test (alpha = 5% threshold)
  Additional information about the measurement:
  2/10: poor 4/10: mediocre 6/10: sufficient 8/10: suitable 10/10: excellent
Image size: comparison of physician satisfaction scores (rated on a scale from 0 to 10) between RU FB and disposable FB | time required to carry out the bronchoscopy (between 5 and 15 minutes)
  A score is given per bronchoscopy (RU FB or disposable FB) All scores are aggregated as an average for FB RU and as an average for disposable FBs The 2 averages obtained are compared by a Student T- test after verification of the application conditions by a Fisher F-test (alpha = 5% threshold)
  Additional information about the measurement:
  2/10: poor 4/10: mediocre 6/10: sufficient 8/10: suitable 10/10: excellent
Reproduction of anatomic reality: comparison of physician satisfaction scores (rated on a scale from 0 to 10) between RU FB and disposable FB | time required to carry out the bronchoscopy (between 5 and 15 minutes)
  A score is given per bronchoscopy (RU FB or disposable FB) All scores are aggregated as an average for FB RU and as an average for disposable FBs The 2 averages obtained are compared by a Student T- test after verification of the application conditions by a Fisher F-test (alpha = 5% threshold)
  Additional information about the measurement:
  2/10: poor 4/10: mediocre 6/10: sufficient 8/10: suitable 10/10: excellent
Suction quality: comparison of physician satisfaction scores (rated on a scale from 0 to 10) between RU FB and disposable FB | time required to carry out the bronchoscopy (between 5 and 15 minutes)
  A score is given per bronchoscopy (RU FB or disposable FB) All scores are aggregated as an average for FB RU and as an average for disposable FBs The 2 averages obtained are compared by a Student T- test after verification of the application conditions by a Fisher F-test (alpha = 5% threshold)
  Additional information about the measurement:
  2/10: poor 4/10: mediocre 6/10: sufficient 8/10: suitable 10/10: excellent

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital, Limoges, Limoges, France

IPD SHARING:
Plan to Share IPD: No